CLINICAL TRIAL: NCT04939155
Title: Measuring the DNA Methylation Effects From COVID-19 Infection and COVID-vaccinations
Brief Title: Methylation Effects of COV-19 Infection and Vaccinations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: TD-ME-001
Record Dates: First submitted 2021-06-14; First posted 2021-06-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients infected with SARS-CoV-2: The first part of this study looks at the methylation patterns in individuals who have a baseline test taken of their DNA methylation patterns in their epigenome and then a follow-up test after they contracted SARS-CoV-2
- Patients who have received an mRNA vaccination: The second part of the study looks at the methylation patterns in individuals who have a baseline test taken of their DNA methylation patterns in their epigenome and then a follow-up test after SARS CoV-2 mRNA vaccine injection.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA vaccine — mRNA vaccine for COVID
  Groups: Patients who have received an mRNA vaccination

SUMMARY:
This is a retrospective non-randomized clinical study of 60 patients total to assess the effects of SARS-CoV-2 infection and the SARS-CoV-2 vaccination. This study will have 2 arms evaluating the epigenomes of patients pre and post-exposure to one of the interventions. The first arm of the study will analyze 40 patients' epigenomes whose DNA methylation was examined pre and post SARS-CoV-2 infection. The second arm of this study is analyzing 20 patients' epigenomes whose DNA methylation was examined pre and post-injection of the SARS-CoV-2 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are healthy individuals and of any sex, ethnicity, and anyone above the age of 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects that are healthy individuals and of any sex, ethnicity, and anyone above the age of 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Methylation age clock testing | Change from baseline after COVID-19 infection
  The DNA clocks that will be used to precisely measure aging is TruAge Biological Age test, which estimates biological age vs. chronological age
Methylation age clock testing | Change from baseline after COVID-19 mRNA vaccination
  The DNA clocks that will be used to precisely measure aging is TruAge Biological Age test, which estimates biological age vs. chronological age

SECONDARY OUTCOMES:
Overall state of health | Change from baseline after COVID-19 infection
  Questionnaire assessing overall health
Overall state of health | Change from baseline after COVID-19 mRNA vaccination
  Questionnaire assessing overall health

CONTACTS AND LOCATIONS:
Locations (1):
- TruDiagnostic, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonek K, Roszkowski L, Massalska M, Maslinski W, Ciechomska M. Biologic Drugs for Rheumatoid Arthritis in the Context of Biosimilars, Genetics, Epigenetics and COVID-19 Treatment. Cells. 2021 Feb 4;10(2):323. doi: 10.3390/cells10020323. PMID 33557301
- [Background] Cao X. COVID-19: immunopathology and its implications for therapy. Nat Rev Immunol. 2020 May;20(5):269-270. doi: 10.1038/s41577-020-0308-3. PMID 32273594
- [Background] Corey L, Mascola JR, Fauci AS, Collins FS. A strategic approach to COVID-19 vaccine R&D. Science. 2020 May 29;368(6494):948-950. doi: 10.1126/science.abc5312. Epub 2020 May 11. No abstract available. PMID 32393526